CLINICAL TRIAL: NCT04174859
Title: Rivaroxaban Treatment Discontinuation Rates in Routine Clinical Practice in Italy in Patients With Non-valvular Atrial Fibrillation
Brief Title: Study Aims to Collect Information in Routine Clinical Practice in Italy About the Number of Patients Suffering From Irregularly Heart Beats Which Are Not Caused by a Heart Valve Problem (Non-valvular Atrial Fibrillation, NVAF) Who Stopped or Changed Rivaroxaban Treatment
Acronym: RITMUS-AF
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 20999
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: Atrial Fibrillation (AF); NVAF
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NVAF patients: Start treatment with rivaroxaban at the discretion of physician.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Treatment dose is following the description of physicians.

SUMMARY:
While it is well known that stopping or changing medication with blood thinners in patients who suffer from non-valvular atrial fibrillation (NVAF) increases the risk of ischemic stroke (a condition which occurs when a vessel supplying blood to the brain is obstructed), bleeding or thromboembolism (a condition that happens when a blood clot forms elsewhere in the body and travels through the blood stream to plug another vessel), limited data are available on the number of NVAF patients and the reasons why NVAF patients in Italy stop or change their treatment with blood thinners to prevent stroke or thromboembolism.

By following the NVAF patients in routine clinical practice in Italy who are treated with rivaroxaban to prevent stroke or systemic embolism researchers want to find out how many NVAF patients and for what reasons NVAF patients stopped or changed rivaroxaban treatment. Study data will be collected through patients' routine visits at their treating doctor over a period of 24 months for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Patient with a diagnosis of NVAF
* New user to rivaroxaban, naïve or non naïve to treatment with oral anticoagulant
* Patient for whom the decision to initiate treatment with rivaroxaban was made as per physician's routine treatment practice for prevention of stroke and non-central nervous system (CNS) systemic embolism
* Signed an informed consent

Exclusion Criteria:

* Patient with heart valve replacement
* Patient is participating in an investigational program with interventions outside of routine clinical practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NVAF patients who are treated with rivaroxaban to prevent stroke or non-CNS systemic embolism. Owing to the observational study design, patients will only be enrolled in the study if the decision to treat with rivaroxaban has been made by the treating physician in advance and independent of study inclusion. The decision to prescribe rivaroxaban is solely at the discretion of the investigator and made in accordance with his/her experience in accordance to SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 812 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Date of start of rivaroxaban treatment | 24 months
Date of stop of rivaroxaban treatment | 24 months
Number of patients who discontinue (i.e: number of discontinuation) from study initiation to end of observation/follow up. | 24 months

SECONDARY OUTCOMES:
Reasons for discontinuation of rivaroxaban therapy | 24 months
  * therapy discontinuation due to adverse event (AE)
  * therapy discontinuation for non AE related reason
  * physician decision
  * patient lost to follow up, no remote contact
  * patient decision (not related to AE)
  * patient is in stable sinus rhythm
  * patient decided to terminate study participation but agreed to further use of data collected so far.
  * patient decided to terminate study participation and refused further use of collected data.
  * Patient died
  * Treatment switch
Reason for dose change of rivaroxaban therapy | 24 months
  * Change in Creatinine Clearance (CrCL)
  * Insufficient therapeutic effect
  * Adverse event
Reason for switch to other therapy | 24 months
  * Ischemic event
  * Bleeding and site of bleeding
  * Adverse drug reaction
  * Drug interaction with other therapies
  * New treatment after switch
Treatment adherence: Self-reported medication adherence measured by the MMAS-8 (Morinsky Scale score) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Italy

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.